CLINICAL TRIAL: NCT05076825
Title: Comparison Of Neurodynamic Sliding Verses Static Stretching On Clinical Outcomes In People With Hamstring Tightness: A Randomized Control Trail
Brief Title: Neurodynamic Sliding Verses Static Stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-UOL-FAHS/761-II/2020
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Healthy Individuals With Hamstring Tightness
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodynamic Sliding (Experimental): participents receive routine physical therapy along with TENS, Hot pack and Neurodynamic Stretching. (For 30 seconds, 3 times per session for 3 alternative days a week & duration of 4 weeks).
  Interventions: Other: Neurodynamic Sliding
- Static Streching (Active Comparator): Participent receive the routine physical therapy treatment that will include TENS, Hot pack and static stretching for 30 seconds and 3 times per session for 3 alternative days a week (duration of 4 weeks).
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Neurodynamic Sliding — Participants supine with their cervical and thoracic spine supported in a forward flexed position. Simultaneous hip and knee flexion will be alternated dynamically with simultaneous hip and knee extension. The therapist will change the arrangement of movement depending on the tissue resistance level.
  Arms: Neurodynamic Sliding
Other: Static Stretching — Participent lying supine, the therapist will passively position the subject into the straight leg raise position without discomfort or pain to the point where resistance to movement will be first felt.
  Arms: Static Streching

SUMMARY:
Hamstring muscle are more likely to shorten among all biarticular muscles of human body. One of the many factors of hamstring tightness is increased tension in the neural structure. Apart from routine stretching techniques, mobilization of nervous system proves to be more effective. There are lot of stretching techniques available but they are more effective after multiple sessions. This study aims to cater the problem of hamstring tightness by neural sliding and static stretching in minimum sessions and compare which technique is more effective in resolving the issue.

DETAILED DESCRIPTION:
Randomized Controlled Trials was used to collect data. Total patients were selected in two group with each 31 subjects. Purposive sampling technique was used. Experimental group will receive routine physical therapy along with TENS, Hot pack and Neurodynamic Stretching. (For 30 seconds, 3 times per session for 3 alternative days a week & duration of 4 weeks). Outcome measure will be the hamstring tightness value angle in degrees, which will be obtained with the help of goniometer after performing active knee extension test and active straight leg raise test

ELIGIBILITY:
Inclusion Criteria:

* People with age ranging between 25 and 35 years.
* Hamstring tightness of twenty degrees
* Incapability to reach seventy degree hip flexion in SLR.

Exclusion Criteria:

* Neurological or orthopedic diseases
* Chronic or acute low back pain, Hamstring injury.
* During last three month, involved in any lower extremity exercise programs.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hamstring flexibility assessed with Active Knee Extension Test | Baseline, 2nd Week, 4th week
  This test is use to measure Hamstring tightness. 0 degree indicates more hamstring flexibility
Change from Baseline in Hamstring flexibility assessed with Straight Leg raise | Baseline, 2nd Week, 4th week
  This test is use to measure hamstring tightness. 90 degree indicates more hamstring flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Mohsin Majeed, Principal Investigator — University of Lahore; Fahad Tanveer, Study Chair — University of Lahore
Locations (1):
- Iqbal Memorial Hospital, Jhang, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No